CLINICAL TRIAL: NCT03594123
Title: A 12-week, Multicenter, Active-treatment Extension Trial to Evaluate the Safety and Tolerability of Brexpiprazole in the Treatment of Subjects With Agitation Associated With Dementia of the Alzheimer's Type
Brief Title: A 12-week Extension Trial to Evaluate the Safety and Tolerability of Brexpiprazole in the Treatment of Subjects With Agitation Associated With Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-201-00182
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer's Disease
Keywords: Agitation
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prior Brexpiprazole (Experimental): Participants who received brexpiprazole in a previous double-blind phase 3 study (Trial 331-14-213 {NCT03548584}), received the same dose of brexpiprazole [2 or 3 milligrams (mg)], once daily (QD), orally, as they received during the previous study, for up to 12 weeks with dose adjustment.
  Interventions: Drug: Brexpiprazole
- Prior Placebo (Experimental): Participants who received placebo in a previous double-blind phase 3 study (Trial 331-14-213 {NCT03548584}), received brexpiprazole following a titration schedule, to gradually increase their dose from 0.5 mg QD, in the starting to 2 or 3 mg QD, orally, for up to 12 weeks with dose adjustment.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — 2 or 3 mg tablet
  Arms: Prior Brexpiprazole
Drug: Brexpiprazole — 0.5 to 3 mg tablet
  Arms: Prior Placebo

SUMMARY:
Active treatment extension study of the 331-14-213 trial, to assess the long-term safety and tolerability of oral brexpiprazole as treatment in adult participants with agitation associated with dementia of the Alzheimer's type (AAD).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have participated in the 331-14-213 study.
* Participants must have an identified caregiver who has contact, at a minimum of 2 hours per day, 4 days per week to describe the participant's symptoms and can observe participant behavior.

Exclusion Criteria:

* Participants with a substantial protocol violation during the course of their participation in the double-blind trial 331-14-213.

Ages: 55 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Shah A, Kalu U, Chen D, Slomkowski M, Hobart M, Such P, Grossberg GT. Brexpiprazole side-effect profile in people with agitation in Alzheimer's dementia: a plain language summary. Curr Med Res Opin. 2026 Jan 14:1-3. doi: 10.1080/03007995.2025.2608578. Online ahead of print. PMID 41533472
- [Derived] Shah A, Estilo A, Sheridan PL, Kalu U, Chen D, Chang D, Slomkowski M, Lee D, Hefting N, Hobart M, Behl S, Such P, Brubaker M, Grossberg GT. Safety and Tolerability of Brexpiprazole in Participants with Agitation Associated with Dementia due to Alzheimer's Disease: Pooled Analysis of Three Randomized Trials and an Extension Trial. CNS Drugs. 2025 Oct;39(10):1011-1023. doi: 10.1007/s40263-025-01200-9. Epub 2025 Jul 19. PMID 40681915
- [Derived] Behl S, Slomkowski M, Chen D, Chang D, Hefting N, Lee D, Shah A, Estilo A, Kalu U, Hobart M. Brexpiprazole for the treatment of agitation associated with dementia due to Alzheimer's disease: A 12-week, active-treatment, extension trial. J Alzheimers Dis. 2024 Nov;102(2):520-529. doi: 10.3233/JAD-240491. Epub 2024 Nov 13. PMID 39534972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 66 sites from 11 October 2018 to 19 September 2022 in the following countries: Bulgaria, Hungary, Serbia, Slovakia, Spain, Ukraine, and the United States.
Pre-assignment Details: Of the 259 participants,163 participants received brexpiprazole and 96 participants received placebo in the parent study 331-14-213. All 259 participants received brexpiprazole in this study. As prespecified in the SAP,data was analyzed based on the treatments (Brexpiprazole or Placebo) received in parent study 331-14-213. Participants received brexpiprazole 2 or 3 mg or placebo in the parent study, data for this study was analyzed and reported in a combined way for brexpiprazole 2 and 3 mg.
Period: Overall Study
Arm/Group | Prior Brexpiprazole | Prior Placebo
Started | 163 | 96
Efficacy Sample: (Efficacy sample comprised of all participants in the safety sample who have a baseline assessment and at least one postbaseline assessment for cohen-mansfield agitation inventory (CMAI) total score.) | 159 | 95
Completed | 142 | 87
Not Completed | 21 | 9
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 8 | 5
Not completed — Site Terminated by Sponsor | 4 | 1
Not completed — Subject Withdrew Consent to Participate | 7 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Other (Not Related to COVID-19) | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized sample comprised of all participants randomized into this trial. As prespecified in the SAP, data was analyzed based on the treatments (Brexpiprazole or Placebo) received in parent study 331-14-213. Participants received brexpiprazole 2 or 3 mg or placebo in the parent study, data for this study was analyzed and reported in a combined way for brexpiprazole 2 and 3 mg.
Groups:
- Prior Brexpiprazole: Participants who received brexpiprazole in a previous double-blind phase 3 study (Trial 331-14-213 {NCT03548584}), received the same dose of brexpiprazole (2 or 3 mg), QD, orally, as they received during the previous study, for up to 12 weeks with dose adjustment.
- Total: Total of all reporting groups
Arm/Group | Prior Brexpiprazole | Prior Placebo | Total
Number analyzed (Participants) | 163 | 96 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (7.9) | 73.4 (73.0) | 74.3 (75.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 46 | 145
  Male | 64 | 50 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 30 | 82
  Not Hispanic or Latino | 111 | 66 | 177
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 154 | 94 | 248
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 15 | 11 | 26
  Hungary | 3 | 2 | 5
  Serbia | 9 | 8 | 17
  Slovakia | 5 | 3 | 8
  Spain | 5 | 3 | 8
  Ukraine | 55 | 31 | 86
  United States | 71 | 38 | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) by Severity
Description: An adverse event (AE) was defined as any untoward medical occurrence in a patient or clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs with an onset date on or after the first dose of brexpiprazole. They are all adverse events that started after start of brexpiprazole; or if the event was continuous from baseline and was worsening, serious, study drug-related, or resulted in death, discontinuation, interruption, or reduction of study therapy.
  Adverse events were graded on a 3-point scale. The intensity of an adverse experience was defined as follows: 1 = Mild: Discomfort noticed, but no disruption to daily activity, 2 = Moderate: Discomfort sufficient to reduce or affect normal daily activity, and 3 = Severe: Inability to work or perform normal daily activity.
Time Frame: From first dose through 30 days after last dose of study drug (Up to approximately Week 16)
Population: Safety Sample comprised of those participants who signed an informed consent form (ICF) for the trial and received at least one dose of brexpiprazole in Trial 331-201-00182. As prespecified in the SAP, data was analyzed based on the treatments (Brexpiprazole or Placebo) received in parent study 331-14-213. Participants received brexpiprazole 2 or 3 mg or placebo in the parent study, data for this study was analyzed and reported in a combined way for brexpiprazole 2 and 3 mg.
Measure: Number; unit: percentage of participants
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 163 | 96
percentage of participants
  Mild | 20.9 | 13.5
  Moderate | 9.2 | 19.8
  Severe | 3.1 | 0

ADVERSE EVENTS:
Time Frame: From first dose through 30 days after last dose of study drug (Up to approximately Week 16)
Description: Safety Sample comprised of those participants who signed an ICF for the trial and received at least one dose of brexpiprazole in Trial 331-201-00182. As prespecified in the SAP, data was analyzed based on the treatments (Brexpiprazole or Placebo) received in parent study 331-14-213. Participants received brexpiprazole 2 or 3 mg or placebo in the parent study, adverse events were analyzed and reported irrespective of the dose, in a combined way for brexpiprazole 2 and 3 mg.
Arm/Group | Prior Brexpiprazole | Prior Placebo
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/96
Serious Adverse Events (participants affected / at risk) | 6/163 | 0/96
Other Adverse Events (participants affected / at risk) | 0/163 | 5/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Brexpiprazole (N=163) | Prior Placebo (N=96)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Brexpiprazole (N=163) | Prior Placebo (N=96)
Nasopharyngitis (Infections and infestations) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03594123/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03594123/SAP_001.pdf